CLINICAL TRIAL: NCT01327404
Title: Myelin, Glia and Depression in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2009-0473; 5R01MH063764 (NIH)
Record Dates: First submitted 2011-03-30; First posted 2011-04-01 (Estimated); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Depression; Diabetes Mellitus
Keywords: Depression; Diabetes Mellitus
MeSH Terms: conditions — Depression; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Depressed: Patients with Major Depressive Disorder
- Diabetic: Patients with Type 2 Diabetes
- Diabetic/Depressed: Patients with both diabetes and major depressive disorder
- Healthy Controls

SUMMARY:
The purpose of the study is to examine the relationship between brain structure and depression in adults aged 30 or older with Diabetes. This relationship is determined using magnetic resonance imaging technology (MRI), a scanner with a magnet that is used to create images of the brain.

DETAILED DESCRIPTION:
Diabetes is a major health problem affecting approximately 18 million Americans. It is a growing crisis that has devastating complications including heart disease, peripheral neuropathy and renal failure. According to a literature review by Gavard et al, the prevalence of major depression in a sample diabetic population in controlled studies was 8.5 to 27.3% (mean prevalence of 14.0%). This was estimated to be up to three times the prevalence of major depression in the general U.S. adult population. Diabetes and major depression are mutual risk factors, with diabetic patients more likely to develop major depression with an odds ratio of 2.5 and depressed patients being more likely to develop type 2 diabetes with an estimated relative risk of 2.2. Depression also has a significant impact on the course of diabetes, leading to higher rates of hyperglycemia and diabetic complications. Depression in patients with diabetes is also associated with poor compliance, decreased quality of life, increased disability and greater health care utilization. A recent 8-year follow-up study of patients with diabetes and depression concluded that the coexistence of these illnesses is associated with a significantly increased risk of death from all causes beyond that due to either depression or diabetes alone. In this study, patients with diabetes and depression had a 1.3-fold increased risk of death from all causes when compared with patients with diabetes alone and a 2-fold increased risk of death when compared with patients with only depression. Reports from a prospective, community-based study in western Australia suggest that the behavioral consequences of depression, including non-compliance with medication and exercise regimens, contribute to increased mortality in these patients.

TRIAL OBJECTIVES AND PURPOSE Specific Aim 1: To study the biophysical properties of the white and gray matter in critical cortical and subcortical regions using magnetization transfer in patients with type 2 diabetes and MDD, non-depressed diabetic controls, patients with unipolar depression without diabetes and nondiabetic healthy controls. The investigators are interested in the separate and cumulative effects of both diabetes and depression on Magnetization Transfer Ratios (MTR) in different brain regions.

Hypothesis: The overarching hypothesis is that both diabetes and depression have the effect of lowering magnetization transfer ratios (MTR) in the anterior cingulate cortex, subcortical nuclei (head of the caudate nucleus and putamen) and the frontal white matter. These effects are cumulative and may not be additive in some regions. Our pilot data suggest that MTR will be lower in these regions in patients with type 2 diabetes (both with and without depression) when compared with healthy controls. In some regions (eg. head of the caudate nucleus - see preliminary data) the investigators anticipate that patients with diabetes and MDD will have the lowest and healthy controls will have the highest MT ratios. The group with unipolar depression without diabetes and the diabetic controls will have MT ratios that fall between these two groups. In other regions of interest, both groups with diabetes will have values significantly different from healthy controls, with patients diagnosed with unipolar depression falling between the healthy and diabetic groups.

Specific Aim 2: To examine levels of glutamate and aspartate (creatine ratios) in two regions involved in the regulation of mood and cognition - the bilateral anterior cingulate cortex and the left subcortical region (the head of the caudate nucleus and the putamen) in patients with type 2 diabetes and our three comparison groups.

Hypothesis: Levels of glutamate and aspartate (creatine ratios) will be lower in patients with combined Type 2 Diabetes and MDD when compared with non-depressed diabetic patients and healthy controls. Our pilot data provide little basis to expect a simple effect of diabetes alone but do not rule out an interaction such that effects are only seen, or are worsened, by the combination of diabetes and depression. The inclusion of a depressed non-diabetic group in the current design will make it possible to evaluate whether the observed effect in the doubly-diagnosed group is best viewed as an effect of depression alone or as an interaction in which diabetes plays a role.

Specific Aim 3: To examine the relationship between regional MTRs and specific cognitive domains in subjects in all four groups.

Hypothesis: There will be direct correlations in all study groups between MT ratios in the subcortical nuclei, anterior cingulate cortex and the dorsolateral white matter and performance on specific cognitive domains, including attention, executive functions, learning and memory and psychomotor processing.

Exploratory Aim 1: In an exploratory manner the investigators will estimate cerebral blood volume, a measure of the cerebral microvasculature, in critical brain regions involved in frontal-subcortical circuitry (anterior cingulate, dorsolateral white, head of the caudate nucleus and the putamen) in subjects in our depressed diabetic group and the three comparison groups using dynamic susceptibility contrast MR imaging (perfusion-weighted MR imaging).

Exploratory Aim 2: A comparison of blood samples from healthy controls, diabetic subjects, depressed subjects and subjects with both depression and diabetes to see if there is evidence of differences in plasma neurotransmitter levels, hypothalamic-pituitary-adrenals (HPA) axis, and immune function between these four subject groups

ELIGIBILITY:
Inclusion Criteria:

* Age: 30 to 80 years old
* Diagnosis of type 2 diabetes
* Diagnosis of major depressive disorder using standard diagnostic and statistical manual (DSM) criteria
* Score of 15 or greater on the 17-item Hamilton Depression rating scale
* Mini Mental Status Exam score of 24 or greater
* No evidence of clinical dementia or any other clinical brain disorder
* Free of psychotropic/psychoactive medications for at least 2 weeks
* First episode of depression diagnosed either after or around the time type 2 diabetes was diagnosed since we are interested in the relationship between the cerebrovascular effect of diabetes and the pathophysiology of major depression

Exclusion Criteria:

* Presence of dementia or any other clinical brain disorder (Parkinson's, Alzheimer's)
* Mini Mental Status Exam score of less than 24
* Unstable medical illness (grade 4 on the Cumulative Illness Rating Scale)
* Presence of any metallic implant that would preclude an MRI scan (pacemaker, etc.)
* Concurrent Axis 1 disorder (schizophrenia, bipolar)
* Use of atypical neuroleptics for the current episode and/or strong clinical suspicion that the diabetes is secondary to the use of atypical neuroleptics;
* Recurrent major depression, operationally defined as two or more, well-characterized episodes of depression, prior to the onset/diagnosis of diabetes
* Seizure disorder
* Stroke/Transient Ischemic Attack
* Central nervous system disorder (multiple sclerosis)
* Trauma to head/Loss of Consciousness
* Claustrophobia
* Eating disorder (anorexia, bulimia)
* Weight of over 350 pounds
* Learning disorder (dyslexia, ADHD)
* Psychosis, panic or anxiety disorder outside the context of depression
* Pregnancy

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of all subject types will be recruited through the general medical, psychiatric, and endocrinology clinics associated with the UIC Medical Center. Patients will be first cleared for participation in the study by their primary physicians. The patient and family will be approached by the PI or another investigator who will explain the research and its goals. We also plan to recruit subjects through flyers and advertisements.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2009-10-19 (Actual); Primary Completion 2014-10-07 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anand Kumar, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois, Chicago, Illinois, United States

REFERENCES:
- [Result] Ajilore O, Narr K, Rosenthal J, Pham D, Hamilton L, Watari K, Elderkin-Thompson V, Darwin C, Toga A, Kumar A. Regional cortical gray matter thickness differences associated with type 2 diabetes and major depression. Psychiatry Res. 2010 Nov 30;184(2):63-70. doi: 10.1016/j.pscychresns.2010.07.003. Epub 2010 Sep 15. PMID 20832254
- [Result] Nguyen TT, Wong TY, Islam FM, Hubbard L, Ajilore O, Haroon E, Darwin C, Esser B, Kumar A. Evidence of early retinal microvascular changes in patients with type 2 diabetes and depression. Psychosom Med. 2010 Jul;72(6):535-8. doi: 10.1097/PSY.0b013e3181da90f4. Epub 2010 Apr 5. PMID 20368470
- [Result] Kumar A, Gupta R, Thomas A, Ajilore O, Hellemann G. Focal subcortical biophysical abnormalities in patients diagnosed with type 2 diabetes and depression. Arch Gen Psychiatry. 2009 Mar;66(3):324-30. doi: 10.1001/archgenpsychiatry.2008.548. PMID 19255382
- [Result] Watari K, Elderkin-Thompson V, Ajilore O, Haroon E, Darwin C, Pham D, Kumar A. Neuroanatomical correlates of executive functioning in depressed adults with type 2 diabetes. J Clin Exp Neuropsychol. 2008 May;30(4):389-97. doi: 10.1080/13803390701440486. PMID 18938677
- See also: Related Info — http://www.psych.uic.edu/